CLINICAL TRIAL: NCT05273086
Title: The Effect of a Sleep Intervention on Sleep Quality in Nursing Students: Study Protocol for a Pilot Randomised Controlled Trial
Brief Title: The Effect of a Sleep Intervention on Sleep Quality in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sleep-UCJC
Record Dates: First submitted 2022-02-03; First posted 2022-03-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Sleep; Healthy Lifestyle

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep intervention program (Experimental): The Sleep Intervention program Group will be subdivided into two groups of 10 participants to receive the sleep quality improvement program. The program consists of 2 sessions of 90 minutes during one week.
  Interventions: Behavioral: Sleep Intervention Group
- Control Group (No Intervention): The control group will continue with their usual routine.

INTERVENTIONS:
Behavioral: Sleep Intervention Group — The intervention group will acquire skills to improve their quality of sleep such as:
  * Acquisition of notions of chronobiology.
  * Location of the nervous structures involved in biological rhythms.
  * Awareness of the existence of three times that direct our biological rhythms, and of the need for them to be synchronized.
  * Self-knowledge of the chronotype and the degree of adjustment of the three times.
  * Knowledge of the variables that determine a good quality of sleep.
  * Applications of chronobiology to the field of nursing. Recommendations for nurses and patients.
  * Self-knowledge of the quality of sleep and the health status of the circadian system.
  Arms: Sleep intervention program

SUMMARY:
The sleep quality in university students is diminished by numerous factors such as alterations in lifestyles, changes, the socio-emotional development or academic performance.The detriment in the quality of sleep can have a negative effects on the quality of life and mental health. It is even a risk factor for cardiovascular diseases. This study is a pilot type clinical trial in which it is intended to implement an intervention to improve the quality of sleep of university nursing students. A randomization of 40 students will be carried out to two treatment groups (intervention n=20 and control n=20). The intervention group will receive two 90-minute sessions during a week where the anatomical structures involved in sleep will be analyzed, workshops will be held to improve the quality of sleep with individual indications after analyzing their rhythms and patterns. The control group will continue with their usual routine.A pre-post evaluation will be carried out on both groups using the Kronowise 3.0 individual wearable bracelet device that measures sleep quality based on general indicators, sleep, wakefulness, internal time, circadian rhythms, temperature, activity, position and light. In addition, information on perceived sleep quality will be collected with the Pittsburgh questionnaire. Sociodemographic data will be collected in the pre measurement for both groups and satisfaction with the program will be collected in the post measurement in the intervention group.

DETAILED DESCRIPTION:
The program consists of 2 sessions of 90 minutes during one week. In the first session, four activities will be carried out: 1) Explanation of the concepts of chronobiology, biological rhythms of the human being, internal clock and synchronizer, and the importance of anatomical structures; 2) Location of the structures mentioned in diagrams and anatomical models of the nervous system; 3) Approach to the concept of chronotype and the existence of three times that affect human circadian rhythms (biological, artificial and social), and how a poor coupling between them leads to a state called chronodisruption; 4) Completion of 2 self-knowledge questionnaires about the sleep pattern. The second session will also consist of four activities: 1) Recommendations on skills to have optimal sleep quality; 2) Carrying out a questionnaire on daytime sleepiness; 3) Applications of the recommendations to the nursing field (work shifts, clinical application in patients); Delivery of the reports to the participants, resolution of questions related to them, and group analysis of the reports of patients with certain circadian pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Students between 18 and 25 years old.
* Students enrolled in the first full Nursing course at Camilo Jose Cela University 2022-23

Exclusion Criteria:

* Previous diagnosis of mental pathology and/or sleep disorders without or with medication (hypnotics, sedatives and melatonin).
* Work activity simultaneous to academic training.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline sleep quality at after intervention. Number of participants who improve their quality of sleep after the intervention evaluated by Kronowise 3.0. | Baseline (before starting the intervention) and post-intervention (3 weeks)
  Kronowise 3.0 wearable wristband individual device. Participants wear the bracelet for 24 hours, 7 days in a row, including weekdays and weekends. Kronowise 3.0 is a multichannel device that continuously records the rhythms of Body Temperature of the skin, Activity (intensity, duration and time), Body Position and light exposure (intensity, type of light, duration and time). All these parameters are registered and combined in a report that indicates the degree of quality of the person's sleep as good, fair or poor. This device is validated as an objective measure of sleep quality equivalent to polysomnography.
Change from baseline perceived sleep quality at after intervention. The Pittsburgh Sleep Quality Index (PSQI) is a vañidated tool that measures the perceived sleep quality. | Baseline (before starting the intervention) and post-intervention (3 weeks)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-assessed questionnaire that measures sleep quality and disturbances over a 1-month time interval. It consists of 19 self-assessed items that are combined into 7 components for a total score of 0 to 21 points (0 indicates good sleep quality and up to 21 points indicates poor quality). The questionnaire has an internal consistency coefficient of 0.81 in the Spanish population.

SECONDARY OUTCOMES:
Date of birth data. Questionnaire developed by researchers. | Baseline (before starting the intervention)
  Date of birth
Toxic habits. Questionnaire developed by researchers. | Baseline (before starting the intervention)
  Data of doses per day regarding the consumption of tobacco, alcohol and drugs.
Physical exercise. The International physical activity questionnaire (IPAQ) is a validated tool to measure the exercise practice of individuals per week. | Baseline (before starting the intervention)
  International physical activity questionnaire (IPAQ) will be used to assess physical activity It is composed of 27-item self-reported physical activity measure collects information about home maintenance activities, gardening, occupational, transportation, free time and sedentary activities. Validity with a Cronbach´s alpha of 0.80. The results are classified into exercise activity levels or categories such as: low, moderate or high. The higher the score, the more level of physical activity they have.
Satisfaction with the intervention. Questionnaire developed by researchers. | Post-intervention (3 weeks).
  Participants from the intervention group will be asked about their satisfaction with the program. It will contains information about their opinion regarding its need, and whether they will be able to recommend it to friends or family, using a Likert scale of 0 to 10 developed by researchers, where 0 is nothing and 10 is completely.
Age in years data. Questionnaire developed by researchers. | Baseline (before starting the intervention)
  Age in years
Gender data. Questionnaire developed by researchers. | Baseline (before starting the intervention)
  Gender
Sleep data. Questionnaire developed by researchers. | Baseline (before starting the intervention)
  sleep coexistence during the study (alone or accompanied)
Anthropometric data. Questionnaire developed by researchers. | Baseline (before starting the intervention)
  Body Mass Index (BMI): height and weight

CONTACTS AND LOCATIONS:
Overall Officials: David Pérez Manchón, Dr, Principal Investigator — Camilo Jose Cela University
Locations (1):
- Cayetana Ruiz Zaldibar, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escobar-Cordoba F, Eslava-Schmalbach J. [Colombian validation of the Pittsburgh Sleep Quality Index]. Rev Neurol. 2005 Feb 1-15;40(3):150-5. Spanish. PMID 15750899
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Brown FC, Buboltz WC Jr, Soper B. Development and evaluation of the Sleep Treatment and Education Program for Students (STEPS). J Am Coll Health. 2006 Jan-Feb;54(4):231-7. doi: 10.3200/JACH.54.4.231-237. PMID 16450848
- [Background] Blazquez A, Martinez-Nicolas A, Salazar FJ, Rol MA, Madrid JA. Wrist skin temperature, motor activity, and body position as determinants of the circadian pattern of blood pressure. Chronobiol Int. 2012 Jul;29(6):747-56. doi: 10.3109/07420528.2012.679328. PMID 22734575
- [Background] Azad MC, Fraser K, Rumana N, Abdullah AF, Shahana N, Hanly PJ, Turin TC. Sleep disturbances among medical students: a global perspective. J Clin Sleep Med. 2015 Jan 15;11(1):69-74. doi: 10.5664/jcsm.4370. PMID 25515274
- [Background] Madrid-Navarro CJ, Puertas Cuesta FJ, Escamilla-Sevilla F, Campos M, Ruiz Abellan F, Rol MA, Madrid JA. Validation of a Device for the Ambulatory Monitoring of Sleep Patterns: A Pilot Study on Parkinson's Disease. Front Neurol. 2019 Apr 11;10:356. doi: 10.3389/fneur.2019.00356. eCollection 2019. PMID 31031690